CLINICAL TRIAL: NCT06894160
Title: Safety and Usability of Adults EXPLORER Exoskeleton in With Neuromuscular Diseases
Brief Title: Safety and Usability of the EXPLORER Exoskeleton in Adults With Neuromuscular Diseases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MarsiBionics (Industry)
Collaborators: Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXP-A-US
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-03

CONDITIONS: Neuromuscular Disorders
Keywords: gait; robotics; neuromuscular disorders; rehabilitation
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults EXPLORER (Experimental): Two sessions with the robotic gait device in patients with neuromuscular diseases.
  Interventions: Device: Adults EXPLORER

INTERVENTIONS:
Device: Adults EXPLORER — Two sessions with the robotic gait device in patients with neuromuscular diseases.

SUMMARY:
Neurodevelopmental disorders frequently result in abnormal development of the Central Nervous System (CNS), often leading to motor impairments such as difficulty in standing and walking. EXPLORER is a robotic exoskeleton for gait rehabilitation, specifically designed for adults aged 18 to 85 with motor disabilities.The aim of this study is to evaluate the safety and usability of the EXPLORER for adults with motor disability.

DETAILED DESCRIPTION:
Neurodevelopmental disorders frequently result in abnormal development of the Central Nervous System (CNS), often leading to motor impairments such as difficulty in standing and walking. EXPLORER is a robotic exoskeleton for gait rehabilitation, specifically designed for adults aged 18 to 85 with motor disabilities. The aim of this study is to evaluate the safety and usability of the EXPLORER for adults with motor disability.

This study will involve testing the gait-assistance exoskeleton in healthy patients during the first phase, and in patients with stroke (ACV), acquired brain injury (DCA), multiple sclerosis (EM), and muscular dystrophy (LM) during the second phase. The study will consist of two phases:

Phase 1: One visit with the device in healthy patients to assess the initial safety and comfort of the device.

Phase 2: A screening visit (S0) followed by two treatment visits with the device (V1-V2) in patients with ACV, DCA, EM, and LM to determine the effectiveness of the device in treating motor impairments caused by these conditions.

The goal of the study is to evaluate the safety and usability of the device in patients with ACV, DCA, EM, and LM, in order to identify potential benefits in improving gait, muscle strength, and overall functionality in this patient group.

ELIGIBILITY:
Inclusion criteria related to the device characteristics:

* Weight < 100 kg.
* Hip width between 30 - 45 cm.
* Distance from the hip joint center to the knee joint center: 36 cm - 50 cm.
* Distance from the knee joint center to the floor: 43.5 cm - 59.5 cm.
* Patients must be able to follow simple instructions.
* MAS < 3 in lower limbs.
* EU shoe size between 36 and 45.
* Absence of pathology affecting movement (only valid for phase 1 of the current study).

Inclusion criteria related to the study:

* Age 18-85 years.
* Diagnosis of stroke (ACV), acquired brain injury (DCA), multiple sclerosis (EM), muscular dystrophy (LM), or cerebral palsy (PC).
* Gait difficulty: those who require assistance to walk using technical aids, assistance, or supervision from others.
* FAC score in participants with DCA, stroke, or MS < 4.
* WISCI II score in participants with MD < 20.

Exclusion Criteria:

* Spasticity (MAS) = 3 in lower limbs.
* Skin alterations in the areas of contact with the device.
* Planned surgical intervention during the study duration.
* Two or more osteoporotic fractures in the lower limbs in the last 2 years.
* Presence of other conditions that cause exercise intolerance (such as uncontrolled hypertension, coronary artery diseases, arrhythmia, congestive heart failure, severe lung disease).
* Surgical operation in the 3 months prior to the start of the study on the limbs and/or spine.
* Psychiatric disorders that interfere with proper use of the device or participation in the study, such as impulsivity or inability to understand simple instructions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | Through study completion, an average of 1 month
  Occurrence of any serious adverse event to the participant or the caregiver
Falls prevalence | Through study completion, an average of 1 month
  Number of falling events occurred from the participant or caregiver
Heart Rate | Through study completion, an average of 1 month
  Beats per minute
Skin integrity | Through study completion, an average of 1 month
  Occurrence of any injury of the skin in the areas of contact and produced by the use of the device
Device usage time | Through study completion, an average of 1 month
  Time using the device
Level of Spasticity | Through study completion, an average of 1 month
  Evaluation of spasticity with Modified Ahsworth Scale
Level of fatigue | Through study completion, an average of 1 month
  Fatigue of both the participant and the therapist, Measured with the Borg scale
Donning and doffing time | Through study completion, an average of 1 month
  Time to don and doff the device to each participant
Level of assistance a participant requires for walking | Through study completion, an average of 1 month
  Measure with FAC scale
Walking ability of individuals with spinal cord injuries | Through study completion, an average of 1 month
  Measure with WISCII (SCI) scale
TUG | Through study completion, an average of 1 month
  The Time Up and Go test is used to assess a participant's mobility and balance
10MWT | Through study completion, an average of 1 month
  The 10-Meter Walk Test is used to assess walking speed by measuring the time taken to walk 10 meters at a comfortable pace.
QUEST 2.0 | at the end of the intervention, an average of 1 month
  Using the Quebec User Evaluation of Satisfaction with Assistive Technology questionnaire administered to the participants' caregivers at the end of the intervention. The QUEST 2.0 scale has 12 items. Each item is rated on a 5-point Likert scale
Blood Pressure | Through study completion, an average of 1 month
  Measure in mmHg
Oxygen Saturation | Through study completion, an average of 1 month
  It analyzes this absorption and calculates the SpO₂

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain